CLINICAL TRIAL: NCT00038129
Title: Study to Prospectively Evaluate Reamed Intramedullary Nails in Tibial Shaft Fractures (SPRINT)
Brief Title: SPRINT - Randomized Trial of Tibial Fracture Fixation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0105M00481; R01AR048529 (NIH); NIAMS-072
Record Dates: First submitted 2002-05-29; First posted 2002-05-30 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Tibial Fracture
MeSH Terms: conditions — Tibial Fractures | interventions — Fracture Fixation, Intramedullary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive reaming of the intramedullary canal prior to insertion of an intramedullary nail.
  Interventions: Procedure: Intramedullary nail implant
- 2 (Experimental): Participants will receive insertion of an intramedullary nail without prior reaming of the intramedullary canal.
  Interventions: Procedure: Intramedullary nail implant

INTERVENTIONS:
Procedure: Intramedullary nail implant — Insertion of an intramedullary nail during tibial fracture fixation with or without prior reaming of the intramedullary canal.

SUMMARY:
The purpose of this study is to determine if there is a difference in the rate of healing of a tibia fracture treated with an intramedullary nail based on whether or not the bone was reamed prior to nail insertion.

DETAILED DESCRIPTION:
Patients with tibia fractures that are amenable to being treated with both a reamed and an unreamed nail will be randomized via telephone to one of the two groups. These patients then will be followed for a year with clinical, as well as subjective, outcome follow-up questionnaires. Time to healing, as well as repeat interventions and adverse events, will be tracked. The rationale for doing a large sample size multi-center trial is the hope that a clear answer to whether or not one of these two methods is significantly better than the other will become apparent and thus aid surgeons in making a more informed operative treatment choice.

ELIGIBILITY:
Inclusion Criteria:

* Fractured tibia requiring fixation using an intramedullary nail

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2002-05; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Necessity for additional operation | Months 6, 9, and 12

SECONDARY OUTCOMES:
Return to work, functional status, and health-related quality of life | Months 6, 9, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Marc F. Swiontkowski, MD, Study Chair — Department of Orthopaedic Surgery, University of Minnesota
Locations (16):
- United States (16):
  - San Francisco General Hospital, San Francisco, California
  - University of Florida - Jacksonville, Jacksonville, Florida
  - Deaconess Hospital, Evansville, Indiana
  - University of Louisville, Louisville, Kentucky
  - Boston Medical Center, Boston, Massachusetts
  - Detroit Receiving Hospital, Detroit, Michigan
  - Regions Hospital, Saint Paul, Minnesota
  - University of Buffalo, Buffalo, New York
  - Jamaica Hospital, Jamaica, New York
  - Wake Medical Center, Raleigh, North Carolina
  - Wake Forest Medical Center, Winston-Salem, North Carolina
  - Metrohealth Medical Center, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Health & Science Univesity, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee
  - Memorial Hermann Hospital, Houston, Texas

REFERENCES:
- [Derived] Schemitsch EH, Kumar A, Heels-Ansdell D, Sprague S, Bhandari M, Guyatt G, Sanders DW, Swiontkowski M, Tornetta P 3rd, Walter S; SPRINT Investigators. Reamed compared with unreamed nailing of tibial shaft fractures: Does the initial method of nail insertion influence outcome in patients requiring reoperations? Can J Surg. 2023 Jul 13;66(4):E384-E389. doi: 10.1503/cjs.012222. Print 2023 Jul-Aug. PMID 37442585
- [Derived] Swiontkowski M, Teague D, Sprague S, Bzovsky S, Heels-Ansdell D, Bhandari M, Schemitsch EH, Sanders DW, Tornetta P, Walter SD; SPRINT Investigators. Impact of centre volume, surgeon volume, surgeon experience and geographic location on reoperation after intramedullary nailing of tibial shaft fractures. Can J Surg. 2021 Jul 5;64(4):E371-E376. doi: 10.1503/cjs.004020. PMID 34222771
- [Derived] Khan JS, Devereaux PJ, LeManach Y, Busse JW. Patient coping and expectations about recovery predict the development of chronic post-surgical pain after traumatic tibial fracture repair. Br J Anaesth. 2016 Sep;117(3):365-70. doi: 10.1093/bja/aew225. PMID 27543531
- [Derived] Busse JW, Bhandari M, Guyatt GH, Heels-Ansdell D, Kulkarni AV, Mandel S, Sanders D, Schemitsch E, Swiontkowski M, Tornetta P 3rd, Wai E, Walter SD; SPRINT Investigators & the Medically Unexplained Syndromes Study Group. Development and validation of an instrument to predict functional recovery in tibial fracture patients: the Somatic Pre-Occupation and Coping (SPOC) questionnaire. J Orthop Trauma. 2012 Jun;26(6):370-8. doi: 10.1097/BOT.0b013e31822421e2. PMID 22011635
- [Derived] SPRINT Investigators; Briel M, Sprague S, Heels-Ansdell D, Guyatt G, Bhandari M, Blackhouse G, Sanders D, Schemitsch E, Swiontkowski M, Tornetta P 3rd, Walter SD, Goeree R. Economic evaluation of reamed versus unreamed intramedullary nailing in patients with closed and open tibial fractures: results from the study to prospectively evaluate reamed intramedullary nails in patients with tibial fractures (SPRINT). Value Health. 2011 Jun;14(4):450-7. doi: 10.1016/j.jval.2010.10.034. Epub 2011 May 25. PMID 21669369
- [Derived] Busse JW, Bhandari M, Guyatt GH, Heels-Ansdell D, Mandel S, Sanders D, Schemitsch E, Swiontkowski M, Tornetta P 3rd, Wai E, Walter SD; SPRINT Investigators. Use of both Short Musculoskeletal Function Assessment questionnaire and Short Form-36 among tibial-fracture patients was redundant. J Clin Epidemiol. 2009 Nov;62(11):1210-7. doi: 10.1016/j.jclinepi.2009.01.014. Epub 2009 Apr 11. PMID 19364637
- [Derived] SPRINT Investigators; Bhandari M, Guyatt G, Tornetta P 3rd, Schemitsch E, Swiontkowski M, Sanders D, Walter SD. Study to prospectively evaluate reamed intramedually nails in patients with tibial fractures (S.P.R.I.N.T.): study rationale and design. BMC Musculoskelet Disord. 2008 Jun 23;9:91. doi: 10.1186/1471-2474-9-91. PMID 18573205